CLINICAL TRIAL: NCT04098744
Title: A Phase II Double Blind, Placebo-controlled, Randomized Trial of Artesunate Vaginal Inserts for the Treatment of Patients With Cervical Intraepithelial Neoplasia (CIN2/3)
Brief Title: Artesunate Vaginal Inserts for the Treatment of Cervical Intraepithelial Neoplasia (CIN2/3)
Acronym: ART-CIN_IIB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Frantz Viral Therapeutics, LLC (Industry)
Collaborators: Amarex Clinical Research (Other); M.D. Anderson Cancer Center (Other); Harris Health System (L.B.J. Hospital) (Unknown); The Cleveland Clinic (Other); University of Michigan (Other); Florida Gynecologic Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-CIN IIB; 2020 0237 (Other: MD Anderson IRB); 20 1148 (Other: CCF IRB)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: CIN 2/3; HPV Infection; Pre-Cancerous Dysplasia; Cervical Dysplasia; HPV Related Disease
Keywords: treatment study; cancer prevention; non-surgical; HPV related disease; CIN; topical treatment; vaginal inserts; artesunate; artemisinin; non-invasive; high risk HPV; vaginal suppository
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia | interventions — artesunic acid; artemisinin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, study team, and sponsor are blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Artesunate vaginal insert (Experimental): Participants will receive three 5-day cycles of artesunate vaginal inserts, 200mg/day, at week 0, week 2, week 4.
  Interventions: Drug: Artesunate vaginal insert
- Placebo vaginal inserts (Placebo Comparator): Participants will receive three 5-day cycles of placebo vaginal inserts, at week 0, week 2, and week 4.
  Interventions: Drug: Placebo vaginal insert

INTERVENTIONS:
Drug: Artesunate vaginal insert — Artesunate formulated as vaginal inserts, 200mg
  Other Names: Artesunic acid; DHA; artemisinin
  Arms: Artesunate vaginal insert
Drug: Placebo vaginal insert — Placebo for artesunate vaginal inserts
  Arms: Placebo vaginal inserts

SUMMARY:
This is a phase II double blind, placebo-controlled, randomized study of Artesunate vaginal inserts for the treatment of women who have cervical high grade intraepithelial neoplasia (CIN2/3).

DETAILED DESCRIPTION:
Eligible participants in this study are randomized 2:1 to receive either artesunate or placebo vaginal inserts for the treatment of CIN2/3. Both groups receive three 5-day cycles of the respective drug, at weeks 0, 2, and 4. Dosing visits can be done as telehealth visits (medication is mailed to the patient's home). Participants are followed after receiving artesunate at weeks 6, 17, and 40. All participants undergo a LEEP procedure at week 17.

Primary Objective: To evaluate the histopathologic response to three 5-day cycles of artesunate vaginal inserts in adult females with biopsy-proven HPV-associated CIN 2/3.

Secondary Objectives:

* To evaluate the safety of artesunate vaginal inserts for the treatment of CIN2/3
* To evaluate the viral clearance after three 5-day cycles of artesunate vaginal inserts in adult females with biopsy-proven HPV-associated CIN 2/3.
* To evaluate viral clearance after three 5-day cycles of artesunate and the LEEP procedure

ELIGIBILITY:
Inclusion Criteria:

* Adult females age ≥ 25 years
* Capable of informed consent
* Any HPV genotype detectable by DNA test/HPV genotyping
* Colposcopically-directed, histologically confirmed tissue diagnosis of cervical high grade squamous intraepithelial lesions (CIN2, CIN3, or CIN2/3)
* Women of childbearing potential agree to use birth control through week17 of the study.
* Weight ≥ 50kg

Exclusion Criteria:

* Pregnant and nursing women
* Active autoimmune disease
* Taking immunosuppressive medication
* HIV seropositivity
* Immunocompromised subjects
* Evidence of concurrent cervical adenocarcinoma in situ
* Concurrent malignancy except for nonmelanoma skin lesions, because treatment for other cancers have systemic effects

Ages: 25 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for women only as it is a treatment for cervical intraepithelial neoplasia (CIN2/3)
Enrollment: 78 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with histologic regression by week 17 | 17 weeks
  Number of participants who undergo histologic regression to cervical intraepithelial neoplasia (CIN) 1 or less by week 17, following three 5-day cycles of artesunate vaginal inserts, as determined by the LEEP histopathologic analysis

SECONDARY OUTCOMES:
Number of participants who have achieved clearance of detectable human papilloma virus (HPV) by week 17 | 17 weeks
  Number of participants who had HPV strains detected at study entry which become undetectable by week 17
Number of participants who have achieved clearance of detectable human papilloma virus (HPV) after three 5-day cycles of artesunate and the LEEP procedure. | 40 weeks
  Number of participants who had HPV strains detected at study entry which become undetectable after three 5-day cycles of artesunate and the LEEP procedure

OTHER OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAE) | 6 weeks
  Number of participants who had adverse events, as defined by CTCAE v5.0, related to the study intervention
Number of participants who withdrew from the study due to TEAEs | 6 weeks
  Number of participants who were withdrawn from the study due to adverse events related to the study drug

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - The Harris Health System (L.B.J Hospital), Houston, Texas
  - University of Texas, M.D. Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No